CLINICAL TRIAL: NCT05372016
Title: A Randomized, Double-Blind and Positive-Controlled Phase 3 Study to Evaluate the Immunogenicity and Safety of the 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha) in Chinese Female Subjects Aged16-26 Years
Brief Title: Evaluate the Immunogenicity and Safety of 9-valent HPV Recombinant Vaccine in Chinese Healthy Females
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Collaborators: Chongqing Bovax Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9-HPV-3002
Record Dates: First submitted 2020-12-27; First posted 2022-05-12 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: HPV Infections; Cervical Cancer; Vulvar Cancer; Vaginal Cancer; CIN1; CIN2; CIN3; VaIN1; VaIN2; VaIN3; Genital Wart; VIN 1; VIN 2; VIN 3; AIS
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) (Experimental): 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) Recombinant Vaccine (Hansenula Polymorpha),0.5mL, three doses, 0,2,6 months
  Interventions: Biological: Experimental: Experimental: 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52, 58)
- GARDASIL ®9 (Active Comparator): GARDASIL®9 (Types 6, 11, 16, 18, 31, 33, 45, 52 and 58) ,0.5mL, three doses, 0,2,6 months
  Interventions: Biological: Active Comparator: GARDASIL ®9

INTERVENTIONS:
Biological: Experimental: Experimental: 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) — 9vHPV vaccine ,0.5mL, three doses, 0,2,6 months
  Arms: Experimental: 9-valent Human Papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52, 58)
Biological: Active Comparator: GARDASIL ®9 — GARDASIL®9 vaccine, 0.5mL, three doses, 0,2,6 months
  Arms: GARDASIL ®9

SUMMARY:
The study will evaluate the immunogenicity and safety of 9-valent HPV recombinant vaccine in Chinese healthy females16 to 26 years of age.

ELIGIBILITY:
Inclusion Criteria:

(If the "*" option is not met during screening, the visit can be rescheduled)

1. Chinese women aged 16-26 who can provide legal identification(If the subject is under 18 years old, proof of legal guardian's identity is also required);
2. The subject agreed to participate in the study, and voluntarily signs the informed consent;for subjects aged 16-18 years, they and their legal guardian(s) are supposed to understand and sign informed consent form together； supposed to understand and sign informed consent form together
3. Subjects are able to understand the study procedures and participate in follow-up according to the study requirements;
4. When the subjects were enrolled, the urine pregnancy test was negative, they were not in the lactation period and had no family planning within 7 months after enrollment.2 weeks before included in the study, effective contraceptive measures has been adopted and agreed to in the first seven months after the study (vaccinations after 1 months ago) continue to adopt effective contraceptive measures (effective contraceptive measures including the pill or condoms, etc ); 5.4. Have an acute illness or an acute episode of a chronic illness within 3 days prior to vaccination or the use of antipyretic, analgesic and antiallergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.);
5. *body temperature <37.3# (underarm body temperature)

Exclusion Criteria:

First dose exclusion criteria(If the "*" option is met during screening, the visit can be rescheduled)

1. Have been vaccinated with commercially available HPV vaccine in the past or planned to be vaccinated with commercially available HPV vaccine during the study period;Or have participated in a clinical trial of the HPV vaccine;
2. Has a history of cervical diseases, such as cervical screening showing abnormal results including CIN or a history of hysterectomy (vaginal or total abdominal hysterectomy) or pelvic radiation therapy. Has a history of genital diseases (such as vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, genital warts, vulvar cancer, vaginal cancer and anal cancer, etc.) or has a previous sexual history (including syphilis, gonorrhea, chancre, venereal lymphatic granuloma, granuloma inguinal);
3. A history of severe allergies requiring medical intervention, such as anaphylactic shock, anaphylactic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc;
4. Subjects present with immune impairment or have been diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases. Long-term immunosuppressive therapy, e.g., long-term (more than 2 weeks) treatment with glucocorticoids (e.g., prednisone or similar drugs);
5. Has been diagnosed with a severe congenital malformation or chronic disease such as Down syndrome, heart disease, liver disease, kidney disease, diabetes, etc., which may interfere with the conduct or completion of the study;
6. Participating in other (drug or vaccine) clinical trials prior to enrollment or planning to participate during the study;
7. Has been diagnosed with an infectious disease, such as tuberculosis, viral hepatitis and/or HIV infection;
8. A history or family history of convulsions, epilepsy, encephalopathy and mental illness;
9. Have contraindications to intramuscular injection, such as having been diagnosed with thrombocytopenia, any coagulation disorder or receiving anticoagulant therapy;
10. Absence of a spleen, functional absence of a spleen, and absence or removal of a spleen in any case;
11. *Have an acute illness or an acute episode of a chronic illness within 3 days prior to vaccination or the use of antipyretic, analgesic and antiallergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.);
12. *Subjects received inactivated or recombinant vaccines within 14 days prior to study enrollment, or attenuated live vaccines within 28 days prior to study enrollment;
13. Subject receives any immunoglobulin or blood product within 3 months prior to the first dose of vaccination;
14. * after questioning, subjects had fever symptoms (subaxillary body temperature ≥37.3#) before the first day of vaccination (within 24 hours before vaccination);
15. Blood pressure on physical examination before the first dose of vaccination was higher than normal or increased (for subjects aged 16-17 year，systolic blood pressure ≥120mmHgand/or diastolic blood pressure ≥80mmHg，for subjects aged 18 year and above，systolic blood pressure ≥140mmHgand/or diastolic blood pressure ≥90mmHg);
16. Subjects may be unable to comply with the study procedure, comply with the agreement, or plan to permanently relocate from the region prior to completion of the study, or may be permanently absent from the region during the scheduled visit;
17. In the opinion of the investigators, the subjects had any other factors that made them unsuitable to participate in the clinical trial.

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
The seroconversion rate of neutralizing antibodies | 30 days after the last dose
  The seroconversion rate of neutralizing antibodies dected after immunization in pre-immune negative subjects from 30 days after the last dose HPV vaccine to HPV 6, 11, 16, 18, 31, 33, 45, 52 , and 58.

SECONDARY OUTCOMES:
Number of subjects with postive antibodies after the whole schedule vaccination from the former negative subjects | 30 days after the last dose
  To evaluate the vaccine immunogenicity is the geometric mean titer from 30 days after the last dose to HPV 6, 11, 16, 18, 31, 33, 45, 52 , and 58.
The level of neutralizing antibody elicited by the vaccine among the subjects with pre-immune positive after the whole schedule vaccination | 30 days after the last dose
  The growth rate of GMTs of anti-HPV 6, 11, 16, 18, 31, 33, 45, 52 and 58 neutralizing antibodies in pre-immune positive subjects from 30 days after immunization
Number of subjects with seroconversion rate (4-fold increase) after the whole schedule vaccination | 30 days after the last dose
  The seroconversion rate (4-fold increase) of anti-HPV 6, 11, 16, 18, 31, 33, 45, 52 and 58 neutralizing antibodies in subjects aged 16-26-year-old from 30 days after immunization
Number of AE within 30 minutes after each dose | 30 mins after each dose
  Adverse events reported within 30 minutes after each dose
Number of SAE within 7days after each dose | day 0 to day 7 after each dose
  Solicited adverse events reported between day 0 to day 7 after each dose
Number of unsolicited adverse events within 30days after each dose | day 0 to day 30 after each dose
  Unsolicited adverse events reported between day 0 to day 30 after each dose
Number of all SAE during the study period | Day 0 to 6 months post vaccination 3
  Serious adverse events reported during the study periodfrom 1st vaccination to the completion of study
Number and rate of pregnancy events | Day 0 to 6 months post vaccination 3
  Pregnant event and pregnant outcome reported during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Guangxi, China